CLINICAL TRIAL: NCT03093961
Title: A Study to Evaluate the Corvia Medical, Inc. IASD® System II to REDUCE Elevated Left Atrial Pressure in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: REDUCE LAP-HFREF TRIAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corvia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1502
Record Dates: First submitted 2017-03-15; First posted 2017-03-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): IASD Implantation
  Interventions: Device: IASD implant

INTERVENTIONS:
Device: IASD implant — Single arm for implant

SUMMARY:
The objective of this pilot study is to evaluate the safety and performance of implanting the IASD® System II in Heart Failure patients with reduced ejection fraction and elevated left sided filling pressures, who remain symptomatic despite Guideline Directed Medical Therapy (GDMT).

DETAILED DESCRIPTION:
The intended clinical indication of the IASD System II is the reduction of elevated LAP in patients with symptomatic heart failure with reduced ejection fraction, despite appropriate medical management. The implant is designed with a center barrel opening that, in the setting of elevated LAP, allows left to right flow. Since many of the symptoms these patients experience are believed to be due to elevated LAP, the IASD System II has the potential to significantly reduce symptoms and improve the quality of life in patients with otherwise limited treatment options.

The study design is a prospective, non-randomized, single-arm feasibility trial. This study will implant up to 10 subjects. The population will include heart failure patients with reduced ejection fraction, and elevated left sided filling pressures, who remain symptomatic despite GDMT, including optimal doses of recommended pharmaceutical treatments, surgical, and device intervention(s) (CRT, AICD, reduction of MRI). After analysis of the 1 month results (including baseline and 1 month Core laboratory echocardiographic and hemodynamic data) of the first 5 implanted patients, a decision will be made to implant an additional 5 patients,

ELIGIBILITY:
Inclusion Criteria:

1. Chronic symptomatic Heart Failure (HF) documented by the following:

   1. New York Heart Association (NYHA) Class III/ambulatory class IV symptoms (Paroxysmal nocturnal dyspnea, Orthopnea, Dyspnea on mild or moderate exertion) at screening visit, and signs (e.g. any rales post cough, Chest x-ray demonstrating pulmonary congestion,) within past 12 months; AND
   2. One hospital admission for which HF was a major component of the hospitalization within the 12 months prior to study entry (transient heart failure in the context of myocardial infarction does not qualify), or one emergency department visit with IV treatment for HF within the 12 months prior to study entry
2. Ongoing stable GDMT for HF (Class I, and IIa recommendations) according to the 2016 ACC/AHA Guidelines for the management of Heart Failure (with no significant changes [>100% increase or 50% decrease], excluding diuretic dose changes for a minimum of 3 months prior to screening), which is expected to be maintained without change for 6 months
3. Age ≥ 18 years old
4. Reduced Left ventricular ejection fraction between 20% and 40% as documented by echocardiography, radio nuclide ventriculography, or MRI within the past 3 months
5. Elevated left atrial pressure with a gradient compared to right atrial pressure (RAP) documented by:

   a. Resting end expiratory PCWP ≥ 18 mmHg, and greater than RAP by ≥ 5 mmHg
6. Subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, as approved by the IRB
7. Subject is willing to comply with clinical investigation procedures and agrees to return for all required follow-up visits, tests, and exams
8. Trans-septal catheterization by femoral vein access is determined to be feasible

Exclusion Criteria:

1. Patients who are not receiving GDMT for specified reasons
2. NT-Pro BNP < 100 pg/mL (if in sinus rhythm), or <300 pg/mL (if in atrial fibrillation); or BNP < 70 pg/mL (if in sinus rhythm), or < 200 pg/mL (if in atrial fibrillation)
3. Myocardial infarction (MI) and/or percutaneous cardiac intervention within past 3 months; CABG in past 3 months, or current indication for coronary revascularization
4. Cardiac Resynchronization Therapy initiated within the past 3 months
5. Automated Implantable Cardioverter Defibrillator (AICD) placed within past 3 months
6. Severe heart failure defined by all of the following:

   1. ACC/AHA/ESC Stage D heart failure, Non-ambulatory NYHA Class IV HF;
   2. Cardiac Index < 2.0 L/min/m2
   3. Requiring inotropic infusion (continuous or intermittent) within the past 3 months.
   4. Listed on transplant waiting list
7. Ability to perform the 6 minute walk Test >600m
8. Known clinically significant un-revascularized coronary artery disease, defined as: epi-cardial coronary artery stenosis associated with angina or other evidence of coronary ischemia.
9. History of stroke, transient ischemic attack (TIA), deep vein thrombosis (DVT), or pulmonary emboli within the past 6 months or recurrent DVT/pulmonary emboli
10. Presence of significant valve disease defined by echocardiography as:

    1. Mitral valve regurgitation defined as grade > 2+ MR
    2. Tricuspid valve regurgitation defined as grade > 2+ TR;
    3. Aortic valve disease defined as ≥ 2+ AR or moderate AS
11. Subject is contraindicated to receive either dual antiplatelet therapy or warfarin analogue; or has a documented coagulopathy
12. Atrial fibrillation with resting HR > 100 BPM
13. Arterial Oxygen saturation < 95% on room air
14. Significant hepatic impairment defined as 3X upper limit of normal of transaminases, total bilirubin, or alkaline phosphatase; Hepatic cirrhosis; Hypoalbuminemia
15. Resting RAP > 14 mmHg
16. Right ventricular dysfunction, defined as

    1. More than mild RV dysfunction as determined by TTE: OR
    2. TAPSE < 1.4 cm: OR
    3. RV volume ≥ LV volume on echo estimate; OR
    4. Evidence of RV dysfunction defined by echo as an RV fractional area change < 35%
17. Evidence of pulmonary hypertension with PVR ≥4 Woods Units
18. Chronic pulmonary disease requiring continuous home oxygen, OR significant chronic pulmonary disease defined as FEV1 <1L.
19. Currently participating in an investigational drug or device study that may interfere with the conduct and outcome of this study.
20. Life expectancy less than 12 months for non-cardiovascular reasons
21. Echocardiographic evidence of intra-cardiac mass, thrombus or vegetation
22. Known or suspected allergy to nickel
23. Women of child bearing potential
24. Currently requiring dialysis; or e-GFR <25ml/min
25. Systolic blood pressure >170 mmHg despite appropriate medical management
26. Subjects with existing or surgically closed (with a patch) Atrial Septal Defects. Subjects with a Patent Foramen Ovale (PFO), who have elevated filling pressure despite the PFO are allowed
27. Subjects on immunosuppression or systemic steroid treatment
28. In the opinion of the investigator, the subject is not an appropriate candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The percent of subjects who experience major adverse cardiac and/or cerebrovascular events (MACCE) | 6 months
  The primary endpoint will be peri-procedural, and 6 months Major Adverse Cardiac and Cerebrovascular Events (MACCE) and systemic embolic events in patients implanted with the IASD.
The percent of subjects who have successful device implantation | Index Procedure
  Deployment at the intended location during the index procedure
The percent of subjects left to right flow through the device | 6 months
  Left to right flow through the device at 6 months as assessed by an echocardiographic core laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Jan Komtebedde, DVM, Study Director — Corvia Medical
Locations (4):
- Mt. Sinai Hospital, New York, New York, United States
- Australia (2):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - St. Vincent Hospital, Sydney
- Homolka Hospital, Prague, Czechia